CLINICAL TRIAL: NCT04562272
Title: Attenuation of Post-infarct Remodeling in Patients With Acute Myocardial Infarction by Left Ventricular Mechanical Unloading Using Impella-CP
Brief Title: Attenuation of Post-infarct LV Remodeling by Mechanical Unloading Using Impella-CP
Acronym: UNLOAD-AMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Marek Sramko, Head of the Department of Acute Cardiology, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15849/20
Record Dates: First submitted 2020-09-20; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Myocardial Infarction; Remodeling, Ventricular; Shock, Cardiogenic
Keywords: ventricular assist device; Impella; unloading
MeSH Terms: conditions — Myocardial Infarction; Ventricular Remodeling; Shock, Cardiogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Mechanical unloading (Active Comparator): Mechanical unloading by Impella-CP for 36-48 hours, on top of the standard treatment
  Interventions: Procedure: LV mechanical unloading by Impella-CP
- Standard care (No Intervention): Standard treatment of AMI after PCI according to guidelines.

INTERVENTIONS:
Procedure: LV mechanical unloading by Impella-CP — The patients will receive Impella-CP for 36-48 hours. The pump speed and LV unloading will be guided by PCWP (Swan-Ganz catheter)
  Other Names: Abiomed Impella-CP
  Arms: Mechanical unloading

SUMMARY:
Patients with anterior wall AMI treated by PCI will undergo, after successful revascularization of the infarct artery, measurement of the left ventricular pressure, and femoral angiogram. Patients with elevated LV pressure and adequate femoral access will be randomized to standard pharmacological treatment of AMI vs. mechanical unloading by Impella-CP (on top of the standard treatment) for 36-48 hours. LV unloading will be guided by measurement of PCWP by Swan-Ganz catheter. On the day 4-7, and at 3 months after the AMI, the patients will undergo SPECT and 3D-echocardiography to assess ventricular remodeling and extent of the post-infarct scar. The patients will be followed for at least 12 months for the occurrence of heart failure and adverse cardiovascular events. The study will test the hypothesis, whether the LV mechanical unloading after PCI will attenuate post-infarct scar and cardiac remodeling.

DETAILED DESCRIPTION:
1. Eligible patients with be screened before PCI
2. The patients with undergo coronary angiography and PCI according to common medical practice
3. At the end of the PCI procedure, after a successful revascularization, a pigtail catheter will be used to measure LV filling pressure and to perform femoral angiography (to evaluate femoral access).
4. Patients fulfilling angiographic and hemodynamic criteria will be randomized 1:1 to standard care vs. mechanical unloading by Impella-CP.
5. The patients will be treated on a CCU with experience with use of Impella-CP.
6. On the CCU, all patients will be monitored by a Swan-Ganz catheter for 48 hours.
7. The pump speed will be adjusted to maintain the lowest tolerated PCWP while avoiding suction events.
8. Mechanical unloading will last 36-48h. Afterwards, the Impella-CP will be explanted.
9. All patients will receive standard pharmacotherapy of AMI, according to the guidelines.
10. Revascularization of significant non-infarct lesions will be performed during the index hospitalization.
11. 3D-echocardiography and Tc-SPECT (D-SPECT) will be performed on the day 5-7 of the index hospitalization. LV phasic volumes and extent of nonperfused myocardium (scar) will be evaluated automatically, using software provided by the vendor.
12. 3D-echocardiography and Tc-SPECT will be repeated at 3 months after the AMI.
13. The patients will be followed by out-patient check-ups every 12 months.

ELIGIBILITY:
Inclusion Criteria:

* large anterior wall AMI with estimated ischemia of <24h
* at risk of the beginning of cardiogenic shock (SCAI A/B)
* blood pressure <160/100 mmHg
* no previous IM based on the patient's history
* no previously known LV systolic dysfunction
* assumed new LV dysfunction documented by ECHO or LVG (LVEF < 45%)
* infarct culprit lesion at the proximal LAD, LMCA or equivalent, with TIMI <= 2 flow
* LV end-diastolic pressure of >= 18 mmHg measured invasively

Exclusion Criteria:

* history of chronic LV dysfunction
* chronic anticoagulation therapy
* the need of IIb/IIIa blockers at the PCI
* inadequate femoral vein access (peripheral artery disease)
* significant valve disease or valve prosthesis
* CPR >5 min before PCI
* LV thrombus
* periprocedural AMI (obliteration of large non-culprit artery during PCI)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in the left ventricular end-systolic volume | LV end-systolic volume measured during the index hospitalization (day 5-7) and at 3 months
  Absolute change in the LVESV measured by SPECT and compared between the groups
Occurrence of LV remodeling | LV end-systolic volume measured during the index hospitalization (day 5-7) and at 3 months
  Occurrence of LV remodeling defined by the increase of LV end-systolic volume >20%
Extent of post-infarct scar | LV scar extent measured during the index hospitalization (day 5-7) and at 3 months
  Extent of post-infarct scar measured by Tc-SPECT and compared between the groups

SECONDARY OUTCOMES:
CV complications | during the first 5 day after AMI
  occurence of TIMI bleeding, hemolysis, thromboembolic events
heart failure | during the first 5 day after AMI
  acute heart failure requiring inotropes or progression of cardiogenic shock

OTHER OUTCOMES:
self-assessed dyspnea | day 1, 2 and 5
  dyspnea reported by the patient on a Likert scale
lung water | day 1, 2 and 5
  assessment of lung water score by ultrasound
maximum hs-TnT, BNP, serum lactate | during the first 5 day after AMI
  diference in hs-TnT, BNP and lactate between the groups

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Clinical and Experimental Medicine (IKEM), Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided